CLINICAL TRIAL: NCT03139721
Title: Medtronic Hancock II® and Mosaic Mitral and Aortic Valves: A Study to Observe the Effects of the Stent Material Change to PEEK Post Approval Study (HAMMOCK PAS)
Brief Title: Medtronic HAMMOCK Post Approval Study
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiac Surgery (Industry)
Responsible Party: Sponsor
Other Study IDs: 1024882DOC
Record Dates: First submitted 2017-04-17; First posted 2017-05-04 (Actual); Results first posted 2024-08-23 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Heart Valve Diseases
MeSH Terms: conditions — Heart Valve Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Primary cohort: Subjects requiring aortic or mitral valve replacement
  Interventions: Device: Mosaic model 305, model 310, and ultra model 305

INTERVENTIONS:
Device: Mosaic model 305, model 310, and ultra model 305 — Aortic or mitral valve replacement
  Other Names: Hancock II model T505, model T510, and ultra model T505

SUMMARY:
This study is being conducted to satisfy the post-CE approval requirement.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who require aortic or mitral valve replacement of their native valve.
2. Subject is geographically stable and willing to return to the implanting site for all follow-up visits.
3. Subject is of legal age to provide informed consent in the country where they enroll in the study.
4. Subject has been adequately informed of risks and requirements of the study and is willing and able to provide informed consent for participation in the clinical study.

Exclusion Criteria:

1. Subject requires concomitant replacement of the aortic and mitral valves.
2. Subject requires a replacement of a previously implanted prosthetic aortic or mitral valve.
3. Subject requires a Bentall procedure for replacement of aortic valve or aortic root.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects requiring aortic or mitral valve replacement of the native valve.
Sampling Method: Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2017-06-19 (Actual); Primary Completion 2019-05-17 (Actual); Study Completion 2021-06-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (4):
  - Franciscan Saint Francis Health, Indianapolis, Indiana
  - ProMedica Toledo Hospital, Toledo, Ohio
  - Saint Joseph Medical Center, Tacoma, Washington
  - Bellin Memorial Hospital, Green Bay, Wisconsin
- Germany (2):
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Deutsches Herzzentrum München Klinik an der TU München, München
- Institute of Cardiology in Warsaw, Warsaw, Poland

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 122 subject were consented to participate. 22 were withdrawn from the study prior to study device implant.
Groups:
- Aortic Valve Replacements: Subjects that received an aortic valve replacement
- Mitral Valve Replacements: Subjects that received a mitral valve replacement
Period: Overall Study
Arm/Group | Aortic Valve Replacements | Mitral Valve Replacements
Started | 89 | 11
Primary Endpoint | 83 | 10
Completed | 68 | 10
Not Completed | 21 | 1

BASELINE CHARACTERISTICS:
Population: Baseline analysis only include subjects implanted with a study valve
Groups:
- Aortic Valve Replacements: Subjects requiring aortic valve replacement
- Mitral Valve Replacements: Subjects requiring mitral valve replacement
- Total: Total of all reporting groups
Arm/Group | Aortic Valve Replacements | Mitral Valve Replacements | Total
Number analyzed (Participants) | 89 | 11 | 100
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Baseline demographics only includes subjects implanted with a study valve.
  Years | 69.6 (7.8) | 69.1 (8.2) | 69.6 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Baseline demographics only include subjects implanted with a study valve
  Participants
    Female | 30 | 4 | 34
    Male | 59 | 7 | 66
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Baseline demographics only include subjects implanted with a study valve
  Participants
    Hispanic or Latino | 0 | 1 | 1
    Not Hispanic or Latino | 75 | 10 | 85
    Unknown or Not Reported | 14 | 0 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Baseline demographics only include subjects implanted with a study valve
  Participants
    American Indian or Alaska Native | 1 | 0 | 1
    Asian | 1 | 0 | 1
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 0 | 1 | 1
    White | 73 | 10 | 83
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 14 | 0 | 14
Region of Enrollment [Number; unit: participants] — Population: Region of enrollment only includes subjects implanted with a study valve
  participants
    United States | 55 | 11 | 66
    Poland | 20 | 0 | 20
    Germany | 14 | 0 | 14
Height [Mean (Standard Deviation); unit: cm] — Population: Baseline demographics only include subjects implanted with a study valve
  cm | 170.3 (9.7) | 170.9 (9.2) | 170.4 (9.6)
Weight [Mean (Standard Deviation); unit: kg] — Population: Baseline demographics only include subjects implanted with a study valve
  kg | 90.2 (19.4) | 88.2 (24.5) | 90.0 (19.9)
Body Surface Area [Mean (Standard Deviation); unit: m^2] — Population: Baseline demographics only include subjects implanted with a study valve
  m^2 | 2.1 (0.3) | 2.0 (0.3) | 2.1 (0.3)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — Population: Baseline demographics only include subjects implanted with a study valve
  kg/m^2 | 31.0 (6.1) | 30.6 (9.8) | 31.0 (6.5)

OUTCOME MEASURES:

1. Primary Outcome: Number of Deaths, Reinterventions, or Explants
Description: Number of deaths, reinterventions, or explants related to the valve
Time Frame: 1-year post implant
Measure: Count of Participants; unit: Participants
Arm/Group | Aortic Valve Replacements | Mitral Valve Replacements
Number analyzed (Participants) | 89 | 11
Participants | 2 | 0

2. Secondary Outcome: Mean Gradient (mmHg)
Description: Measured by echocardiogram via Echo Core Lab
Time Frame: 1-year post implant
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Aortic Valve Replacements | Mitral Valve Replacements
Number analyzed (Participants) | 81 | 10
mmHg | 14.3 (5.1) | 4.6 (1.8)

3. Secondary Outcome: Peak Gradient (mmHg)
Description: Measured by echocardiogram via Echo Core Lab
Time Frame: 1-year post implant
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Aortic Valve Replacements | Mitral Valve Replacements
Number analyzed (Participants) | 81 | 10
mmHg | 25.6 (9.2) | 11.2 (4.1)

4. Secondary Outcome: Effective Orifice Area (EOA)
Description: Measured by echocardiogram via Echo Core Lab
Time Frame: 1-year post implant
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | Aortic Valve Replacements | Mitral Valve Replacements
Number analyzed (Participants) | 72 | 10
cm^2 | 1.41 (0.37) | 1.35 (0.43)

5. Secondary Outcome: Effective Orifice Area Index (EOAi)
Description: EOA Measured by echocardiogram via Echo Core Lab/Body Surface Area
Time Frame: 1-year post implant
Measure: Mean (Standard Deviation); unit: cm^2/m^2
Arm/Group | Aortic Valve Replacements | Mitral Valve Replacements
Number analyzed (Participants) | 72 | 10
cm^2/m^2 | 0.71 (0.18) | 0.70 (0.24)

6. Secondary Outcome: Cardiac Output
Description: Measured by echocardiogram via Echo Core Lab
Time Frame: 1-year post implant
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Aortic Valve Replacements | Mitral Valve Replacements
Number analyzed (Participants) | 70 | 10
L/min | 4.7 (1.1) | 4.1 (1.2)

7. Secondary Outcome: Cardiac Index
Description: Cardiac Output Measured by echocardiogram via Echo Core Lab/Body Surface Area
Time Frame: 1-year post implant
Measure: Mean (Standard Deviation); unit: L/min/m^2
Arm/Group | Aortic Valve Replacements | Mitral Valve Replacements
Number analyzed (Participants) | 70 | 10
L/min/m^2 | 2.4 (0.5) | 2.1 (0.4)

8. Secondary Outcome: Performance Index
Description: The performance index is a measure of how effectively the external dimension of the valve is used to provide forward flow, normalized to the valve size. It is defined as effective orifice area divided by the tissue annulus area, where the tissue annulus area is calculated from the prosthetic valve size.
Time Frame: 1-year post implant
Measure: Mean (Standard Deviation); unit: Units do not exist
Arm/Group | Aortic Valve Replacements | Mitral Valve Replacements
Number analyzed (Participants) | 72 | 10
Units do not exist | 0.4 (0.1) | 0.2 (0.1)

9. Secondary Outcome: Transvalvular Regurgitation
Description: Measured by echocardiogram via Echo Core Lab
Time Frame: 1-year post implant
Measure: Count of Participants; unit: Participants
Arm/Group | Aortic Valve Replacements | Mitral Valve Replacements
Number analyzed (Participants) | 81 | 10
Participants
  None | 67 | 7
  Trace | 6 | 2
  Mild | 1 | 1
  Moderate | 0 | 0
  Moderate to Severe | 0 | 0
  Severe | 0 | 0
  Not recorded/unable to assess | 7 | 0

10. Secondary Outcome: Paravalvular Regurgitation
Description: Measured by echocardiogram via Echo Core Lab
Time Frame: 1-year post implant
Measure: Count of Participants; unit: Participants
Arm/Group | Aortic Valve Replacements | Mitral Valve Replacements
Number analyzed (Participants) | 81 | 10
Participants
  None | 64 | 9
  Trace | 1 | 0
  Mild | 6 | 0
  Moderate | 3 | 0
  Moderate to Severe | 0 | 0
  Severe | 0 | 0
  Not recorded/unable to assess | 7 | 1

11. Secondary Outcome: Total Regurgitation
Description: Measured by echocardiogram via Echo Core Lab
Time Frame: 1-year post implant
Measure: Count of Participants; unit: Participants
Arm/Group | Aortic Valve Replacements | Mitral Valve Replacements
Number analyzed (Participants) | 81 | 10
Participants
  None | 58 | 6
  Trace | 7 | 2
  Mild | 9 | 1
  Moderate | 3 | 0
  Moderate to Severe | 0 | 0
  Severe | 0 | 0
  Not recorded/unable to assess | 4 | 1

12. Secondary Outcome: New York Heart Association (NYHA) Classification
Description: Measure Description: Cardiac Disease with Functional Classes (lower value is more desirable than higher value) I - No limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation or shortness of breath.
  II - Slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, shortness of breath or chest pain.
  III - Marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes fatigue, palpitation, shortness of breath or chest pain.
  IV - Symptoms of heart failure at rest. Any physical activity causes further discomfort.
Time Frame: 1-year post implant
Measure: Count of Participants; unit: Participants
Arm/Group | Aortic Valve Replacements | Mitral Valve Replacements
Number analyzed (Participants) | 75 | 10
Participants
  NYHA I | 51 | 8
  NYHA II | 21 | 2
  NYHA III | 3 | 0
  NYHA IV | 0 | 0

13. Primary Outcome: Number of Deaths, Reinterventions, or Explants
Description: Number of deaths, reinterventions, or explants related to the valve
Time Frame: 3-years post implant
Measure: Count of Participants; unit: Participants
Arm/Group | Aortic Valve Replacements | Mitral Valve Replacements
Number analyzed (Participants) | 89 | 11
Participants | 2 | 0

14. Secondary Outcome: Mean Gradient
Description: Measured by echocardiogram via Echo Core Lab
Time Frame: 3-years post implant
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Aortic Valve Replacements | Mitral Valve Replacements
Number analyzed (Participants) | 59 | 6
mmHg | 14.3 (4.4) | 5.0 (1.3)

15. Secondary Outcome: Peak Gradient
Description: Measured by echocardiogram via Echo Core Lab
Time Frame: 3-years post implant
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Aortic Valve Replacements | Mitral Valve Replacements
Number analyzed (Participants) | 59 | 6
mmHg | 26.5 (8.3) | 11.3 (3.4)

16. Secondary Outcome: Effective Orifice Area (EOA)
Description: Measured by echocardiogram via Echo Core Lab
Time Frame: 3-years post implant
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | Aortic Valve Replacements | Mitral Valve Replacements
Number analyzed (Participants) | 48 | 6
cm^2 | 1.41 (0.32) | 1.26 (0.47)

17. Secondary Outcome: Effective Orifice Area Index (EOAi)
Description: EOA Measured by echocardiogram via Echo Core Lab/Body Surface Area
Time Frame: 3-years post implant
Measure: Mean (Standard Deviation); unit: cm^2/m^2
Arm/Group | Aortic Valve Replacements | Mitral Valve Replacements
Number analyzed (Participants) | 48 | 6
cm^2/m^2 | 0.71 (0.14) | 0.63 (0.22)

18. Secondary Outcome: Cardiac Output
Description: Measure by echocardiogram via Echo Core Lab
Time Frame: 3-years post implant
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Aortic Valve Replacements | Mitral Valve Replacements
Number analyzed (Participants) | 49 | 7
L/min | 4.7 (1.0) | 3.6 (0.7)

19. Secondary Outcome: Cardiac Index
Description: Cardiac output measured by echocardiogram via Echo Core Lab/Body Surface Area
Time Frame: 3-years post implant
Measure: Mean (Standard Deviation); unit: L/min/m^2
Arm/Group | Aortic Valve Replacements | Mitral Valve Replacements
Number analyzed (Participants) | 49 | 7
L/min/m^2 | 2.4 (0.5) | 1.8 (0.3)

20. Secondary Outcome: Performance Index
Description: as for outcome 8
Time Frame: 3-years post implant
Measure: Mean (Standard Deviation); unit: Units do not exist
Arm/Group | Aortic Valve Replacements | Mitral Valve Replacements
Number analyzed (Participants) | 48 | 6
Units do not exist | 0.4 (0.1) | 0.2 (0.1)

21. Secondary Outcome: Transvalvular Regurgitation
Description: Measured by echocardiogram via Echo Core Lab
Time Frame: 3-years post implant
Measure: Count of Participants; unit: Participants
Arm/Group | Aortic Valve Replacements | Mitral Valve Replacements
Number analyzed (Participants) | 59 | 9
Participants
  None | 50 | 4
  Trace | 1 | 4
  Mild | 1 | 1
  Moderate | 0 | 0
  Moderate to Severe | 0 | 0
  Severe | 0 | 0
  Not recorded/unable to assess | 7 | 0

22. Secondary Outcome: Paravalvular Regurgitation
Description: Measured by echocardiogram via Echo Core Lab
Time Frame: 3-years post implant
Measure: Count of Participants; unit: Participants
Arm/Group | Aortic Valve Replacements | Mitral Valve Replacements
Number analyzed (Participants) | 59 | 9
Participants
  None | 46 | 9
  Trace | 1 | 0
  Mild | 4 | 0
  Moderate | 1 | 0
  Moderate to Severe | 0 | 0
  Severe | 0 | 0
  Not recorded/Unable to assess | 7 | 0

23. Secondary Outcome: Total Regurgitation
Description: Measured by echocardiogram via Echo Core Lab
Time Frame: 3-years post implant
Measure: Count of Participants; unit: Participants
Arm/Group | Aortic Valve Replacements | Mitral Valve Replacements
Number analyzed (Participants) | 59 | 9
Participants
  None | 44 | 4
  Trace | 3 | 4
  Mild | 6 | 1
  Moderate | 1 | 0
  Moderate to Severe | 2 | 0
  Severe | 0 | 0
  Not recorded/Unable to assess | 3 | 0

24. Secondary Outcome: New York Heart Association (NYHA) Classification
Description: as for outcome 12
Time Frame: 3-years post implant
Measure: Count of Participants; unit: Participants
Arm/Group | Aortic Valve Replacements | Mitral Valve Replacements
Number analyzed (Participants) | 66 | 9
Participants
  NYHA I | 51 | 7
  NYHA II | 14 | 1
  NYHA III | 1 | 1
  NYHA IV | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Aortic Valve Replacements | Mitral Valve Replacements
All-Cause Mortality (participants affected / at risk) | 8/89 | 1/11
Serious Adverse Events (participants affected / at risk) | 55/89 | 7/11
Other Adverse Events (participants affected / at risk) | 52/89 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aortic Valve Replacements (N=89) | Mitral Valve Replacements (N=11)
Anaemia (Blood and lymphatic system disorders) | 4 (5) | 0 (0)
Blood Loss Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Acute Myocardial Infarction (Cardiac disorders) | 2 (2) | 0 (0)
Arrhythmia Supraventricular (Cardiac disorders) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 5 (5) | 1 (1)
Atrial Rupture (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular Block Complete (Cardiac disorders) | 2 (2) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac Arrest (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac Failure Acute (Cardiac disorders) | 4 (4) | 0 (0)
Cardiac Failure Congestive (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac Tamponade (Cardiac disorders) | 2 (2) | 0 (0)
Cardiogenic Shock (Cardiac disorders) | 1 (1) | 1 (1)
Coronary Artery Disease (Cardiac disorders) | 1 (1) | 1 (1)
Ischaemic Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Low Cardiac Output Syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial Effusion (Cardiac disorders) | 2 (2) | 0 (0)
Pericardial Haemorrhage (Cardiac disorders) | 2 (2) | 0 (0)
Right Ventricular Dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Sinus Node Dysfunction (Cardiac disorders) | 4 (4) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Tricuspid Valve Incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular Asystole (Cardiac disorders) | 0 (0) | 1 (1)
Retinal Artery Occlusion (Eye disorders) | 1 (1) | 0 (0)
Abdominal Compartment Syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Alcoholic Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal Hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal Stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis Acute (Gastrointestinal disorders) | 1 (1) | 1 (1)
Umbilical Hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Multiple Organ Dysfunction Syndrome (General disorders) | 2 (2) | 0 (0)
Cholecystitis Acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Abscess Limb (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 2 (2) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 1 (2)
Covid-19 (Infections and infestations) | 1 (1) | 0 (0)
Endocarditis (Infections and infestations) | 1 (1) | 1 (1)
Endocarditis Enterococcal (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 2 (2)
Postoperative Wound Infection (Infections and infestations) | 2 (3) | 0 (0)
Pulmonary Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal Abscess (Infections and infestations) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Wound Infection (Infections and infestations) | 2 (2) | 0 (0)
Ankle Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cardiac Vein Perforation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Carotid Artery Restenosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament Rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postpericardiotomy Syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural Pneumothorax (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Tibia Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ulna Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular Pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound Dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Human Metapneumovirus Test (Investigations) | 1 (1) | 0 (0)
Calciphylaxis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Compartment Syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Adenocarcinoma Of Colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Invasive Ductal Breast Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Carotid Artery Stenosis (Nervous system disorders) | 1 (1) | 2 (2)
Cerebral Infarction (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Hepatic Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic Stroke (Nervous system disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Transient Ischaemic Attack (Nervous system disorders) | 1 (1) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 5 (5) | 1 (1)
End Stage Renal Disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Oliguria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal Impairment (Renal and urinary disorders) | 2 (2) | 0 (0)
Urinary Bladder Haemorrhage (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary Retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Scrotal Oedema (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (2)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 0 (0)
Pulmonary Air Leakage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Thoracic Cavity Drainage (Surgical and medical procedures) | 1 (1) | 0 (0)
Aortic Aneurysm (Vascular disorders) | 2 (2) | 0 (0)
Aortic Dissection (Vascular disorders) | 2 (2) | 0 (0)
Aortic Stenosis (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 0 (0)
Jugular Vein Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Peripheral Arterial Occlusive Disease (Vascular disorders) | 1 (1) | 0 (0)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aortic Valve Replacements (N=89) | Mitral Valve Replacements (N=11)
Anaemia (Blood and lymphatic system disorders) | 18 (18) | 6 (6)
Blood Loss Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 18 (19) | 7 (7)
Thrombocytopenia (Blood and lymphatic system disorders) | 13 (13) | 10 (10)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 21 (21) | 4 (4)
Atrial Flutter (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular Block First Degree (Cardiac disorders) | 0 (0) | 4 (4)
Bradycardia (Cardiac disorders) | 0 (0) | 2 (2)
Bundle Branch Block Left (Cardiac disorders) | 0 (0) | 1 (1)
Bundle Branch Block Right (Cardiac disorders) | 0 (0) | 1 (1)
Nodal Rhythm (Cardiac disorders) | 0 (0) | 4 (4)
Pericardial Effusion (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial Rub (Cardiac disorders) | 0 (0) | 3 (3)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Sinus Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular Extrasystoles (Cardiac disorders) | 0 (0) | 3 (3)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Vision Blurred (Eye disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 5 (5) | 5 (5)
Nausea (Gastrointestinal disorders) | 0 (0) | 7 (7)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 5 (5) | 1 (1)
Impaired Healing (General disorders) | 0 (0) | 1 (1)
Oedema Peripheral (General disorders) | 7 (7) | 0 (0)
Physical Deconditioning (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Anaemia Postoperative (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Depression Postoperative (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Face Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood Creatinine Increased (Investigations) | 0 (0) | 1 (1)
Blood Urea Nitrogen/Creatinine Ratio Increased (Investigations) | 0 (0) | 1 (1)
Cardiac Index Decreased (Investigations) | 0 (0) | 1 (1)
Prothrombin Time Ratio Increased (Investigations) | 0 (0) | 1 (1)
Electrolyte Imbalance (Metabolism and nutrition disorders) | 12 (12) | 10 (10)
Fluid Overload (Metabolism and nutrition disorders) | 6 (7) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 12 (12) | 10 (10)
Hypervolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Iron Deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Vitamin B12 Deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 3 (3)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Confusional State (Psychiatric disorders) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 6 (6) | 4 (4)
Urinary Retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 5 (5)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary Air Leakage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pulmonary Vascular Disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 8 (8)
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Subcutaneous Emphysema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 8 (8) | 6 (6)
Hypotension (Vascular disorders) | 8 (9) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI is restricted to publish results until the Sponsor has published the results.

DOCUMENTS (2):
  • Study Protocol (2017-11-13): https://cdn.clinicaltrials.gov/large-docs/21/NCT03139721/Prot_000.pdf
  • Statistical Analysis Plan (2017-04-14): https://cdn.clinicaltrials.gov/large-docs/21/NCT03139721/SAP_001.pdf